CLINICAL TRIAL: NCT05349786
Title: The Effect of the Physical Activity Program on Quality of Life, Functional Capacity and Mortality Risk Level in Individuals With Heart Failure
Brief Title: Physical Activity Program on Clinical Output in Heart Failure
Acronym: Heartfailu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Arzu Senturk, Principal Investigator, Research Assistant (RN, MSN, PhD), Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NOHU- Cardiac Nursing
Record Dates: First submitted 2022-04-16; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure; Nursing Caries
Keywords: Heart failure; Physical activity; Functional capacity; Quality of life; NT-proBNP; Mortality risk level
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A physical activity program lasting at least 30 minutes each session was applied to HF patients in the intervention group, three days a week for three months. A pedometer was used to visualize the walking performed in the physical activity program and to record reliably. Weekly phone calls and monthly home visits were made to the patients in order to determine the continuation of the medical treatment and walking program used by the patients, to increase their motivation and to detect or intervene in any situation related to the walking program.
  Interventions: Other: Physical activity program
- Non-Intervention Group (No Intervention): The individuals in the control group, were pre-tested, evaluated at the first, second, and third months, and followed up in the process without any intervention. Patients were reminded that they should continue their routine medical treatment and not start any physical activity program.

INTERVENTIONS:
Other: Physical activity program — A physical activity program lasting at least 30 minutes each session was applied to HF patients in the intervention group, three days a week for three months. A pedometer was used to visualize the walking performed in the physical activity program and to record reliably. After the data obtained in the pre-test, the pedometers, which were calibrated and checked by the researchers, were delivered to the patients. At the end of each day of walking with pedometer monitoring, they were asked to record data such as the number of steps, walking hour, walking time, distance and complaints encountered during walking on the walking monitoring chart given to the patient by the researchers. Weekly phone calls and monthly home visits were made to the patients in order to determine the continuation of the medical treatment and walking program used by the patients, to increase their motivation and to detect or intervene in any situation related to the walking program.
  Arms: Intervention Group

SUMMARY:
Background: This study was carried out to determine the effect of physical activity program applied to individuals with heart failure on quality of life, functional capacity and mortality risk level.

Objective: The study, which was conducted as a randomized controlled experimental study, was completed with a total of 40 HF patients, 20 of whom were interventions and 20 were controls. A physical activity program lasting at least 30 minutes each session was applied to HF patients in the intervention group, three days a week for three months, and the walks of the patients were followed by a pedometer.

DETAILED DESCRIPTION:
Background: This study was carried out to determine the effect of physical activity program applied to individuals with heart failure on quality of life, functional capacity and mortality risk level.

Objective: The study, which was conducted as a randomized controlled experimental study, was completed with a total of 40 HF patients, 20 of whom were interventions and 20 were controls. A physical activity program lasting at least 30 minutes each session was applied to HF patients in the intervention group, three days a week for three months, and the walks of the patients were followed by a pedometer. At the same time, a monthly home visit and weekly phone call were made to the patients. No intervention was applied to the patients in the control group, apart from weekly phone calls. All patients were receiving optimal stable HF therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Class I, II, III according to NYHA classification,
* Without any diagnosis of musculoskeletal deformity or disease that may prevent them from doing physical activity,
* Hypertension stage 1 and 2,
* Stable chronic disease processes such as diabetes,
* Patients whose treatment for these diagnoses has not been changed in the last month,
* Dyspnea status less than 4-5 degrees according to the Modified Borg Scale,
* Cognitive competence,
* At least primary school graduates

Exclusion Criteria:

* Known and diagnosed moderate or severe mitral/aortic regurgitation, hypertrophic obstructive cardiomyopathy, uncontrollable arrhythmia (atrial fibrillation etc.), bundle branch block on ECG,
* Acute myocardial infarction in the last three months,
* Unstable angina pectoris, pacemaker, valve surgery, coronary artery bypass surgery history, newly diagnosed or suspected thromboembolic event,
* Diagnosed with cerebrovascular and peripheral vascular insufficiency, other chronic diseases (such as chronic obstructive pulmonary disease, chronic kidney failure, pulmonary emphysema, rheumatic valve disease, cancer diagnosis),
* Chronic fatigue syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Quality of Life Level | Change from baseline scores at the first month, second month, third month scores
  Quality of life level were evaluated with the Minnesota Living with Heart Failure Questionnaire. Minnesota Living with Heart Failure Questionnaire was developed by Rector et al. to measure the quality of life in patients with heart failure. The total score of the scale, which has two sub-dimensions as "physical function" and "emotional", varies between 0 and 105. A low score indicates good quality of life, and a high score indicates poor quality of life.
Functional Capacity Level | Change from baseline scores at the first month, second month, third month scores
  Functional capacity level was evaluated with the International Physical Activity Questionnaire-Short Form and 6-Min Walking Test. International Physical Activity Questionnaire- Short Form developed by Craig et al. evaluates the duration of physical activity in the last seven days and the time spent sitting per day without moving. The energy required for each activity in the IPAQ is calculated with the metabolic equivalent-minute score according to the activity type or intensity. Functional capacity was evaluated with 6MWT according to the criteria of the "American Thoracic Society" guideline and the 6MWT distance reached at the end of the test was recorded in meters (m). In the study, the blood pressure of individuals was measured before and after 6MWT. Oxygen saturation and heart rate measurements were made and recorded with a portable pulse oximeter.
Mortality Risk Level | Change from baseline scores at the first month, second month, third month scores
  Mortality risk level was evaluated with Meta-Analysis Global Group in Chronic Heart Failure scores. To predict one- and three-year mortality in HF, with MAGGIC, Pocock et al. (2013) analyzed 30 cohort studies with a large number of patients, and they developed a risk scoring database based on HF risk factors. MAGGIC risk scoring results, provides a preliminary assessment in determining the one-year mortality in HF patients. In our study, the MAGGIC scores, which were obtained by taking the scores related to the initial and final follow-up, were compared. NT-proBNP serum concentration measurements, especially ventricular ischemic injury, have an important place in the prediction of mortality. In our study, serum NT-proBNP level was investigated to determine the diagnosis and prognosis of HF, to determine the functional capacity and the relationship between MAGGIC risk scoring and mortality risk.
Severity of Fatigue | Change from baseline scores at the first month, second month, third month scores
  Fatigue Severity Scale used to evaluate the severity of fatigue in the last month was developed by Krupp in 1989. The low total score of the scale with a cut-off value of 4 and above for pathological fatigue indicates low fatigue.

SECONDARY OUTCOMES:
Echocardiographic Evaluation | Change from baseline scores at the end of third month
  There is a LVEF finding as an Echo finding made by the physician to be used in the MAGGIC scoring calculation. Considering that Echo evaluation may vary according to the physician's follow-up, it was ensured that the EF levels of the individuals were performed by the operator who performed the initial follow-up.
Cardiac Enzymes of Laboratory Investigation | Change from baseline scores at the end of third month
  The biochemical variables that may accompany the cause and functional classification of HF were taken from the file information. Among the biochemical values, cardiac enzymes troponin and LDH and NT-proBNP levels were examined.
HbA1c of Laboratory Investigation | Change from baseline scores at the end of third month
  The HbA1c within biochemical variables that may accompany the cause and functional classification of HF were taken from the file information. Among the biochemical values, HbA1c levels were investigated in order to evaluate the regulated status of individuals with diabetes mellitus and the effect of physical activity program.
Body Composition | Change from baseline scores at the first month, second month, third month scores
  In order to evaluate the effect of the physical activity program on the body analysis results, measurement parameter data and body mass index composition (BMI in kg/m^2) (e.g. body weight, body mass index, body fat rate, body muscle mass, body water rate, basal metabolic rate) were obtained from the individuals using a body analysis scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Arzu ŞENTÜRK, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleg JL, Cooper LS, Borlaug BA, Haykowsky MJ, Kraus WE, Levine BD, Pfeffer MA, Pina IL, Poole DC, Reeves GR, Whellan DJ, Kitzman DW; National Heart, Lung, and Blood Institute Working Group. Exercise training as therapy for heart failure: current status and future directions. Circ Heart Fail. 2015 Jan;8(1):209-20. doi: 10.1161/CIRCHEARTFAILURE.113.001420. No abstract available. PMID 25605639
- [Background] Hassanpour Dehkordi A, Khaledi Far A. Effect of exercise training on the quality of life and echocardiography parameter of systolic function in patients with chronic heart failure: a randomized trial. Asian J Sports Med. 2015 Mar;6(1):e22643. doi: 10.5812/asjsm.22643. Epub 2015 Mar 20. PMID 25883771
- [Background] Vetrovsky T, Siranec M, Parenica J, Griva M, Stastny J, Precek J, Pelouch R, Bunc V, Linhart A, Belohlavek J. Effect of a 6-month pedometer-based walking intervention on functional capacity in patients with chronic heart failure with reduced (HFrEF) and with preserved (HFpEF) ejection fraction: study protocol for two multicenter randomized controlled trials. J Transl Med. 2017 Jul 3;15(1):153. doi: 10.1186/s12967-017-1257-x. PMID 28673328
- [Background] Teng HC, Yeh ML, Wang MH. Walking with controlled breathing improves exercise tolerance, anxiety, and quality of life in heart failure patients: A randomized controlled trial. Eur J Cardiovasc Nurs. 2018 Dec;17(8):717-727. doi: 10.1177/1474515118778453. Epub 2018 May 18. PMID 29775076
- [Background] van Tol BA, Huijsmans RJ, Kroon DW, Schothorst M, Kwakkel G. Effects of exercise training on cardiac performance, exercise capacity and quality of life in patients with heart failure: a meta-analysis. Eur J Heart Fail. 2006 Dec;8(8):841-50. doi: 10.1016/j.ejheart.2006.02.013. Epub 2006 May 18. PMID 16713337
- [Background] Nolte K, Herrmann-Lingen C, Wachter R, Gelbrich G, Dungen HD, Duvinage A, Hoischen N, von Oehsen K, Schwarz S, Hasenfuss G, Halle M, Pieske B, Edelmann F. Effects of exercise training on different quality of life dimensions in heart failure with preserved ejection fraction: the Ex-DHF-P trial. Eur J Prev Cardiol. 2015 May;22(5):582-93. doi: 10.1177/2047487314526071. Epub 2014 Mar 13. PMID 24627449
- [Background] Maldonado-Martin S, Brubaker PH, Eggebeen J, Stewart KP, Kitzman DW. Association Between 6-Minute Walk Test Distance and Objective Variables of Functional Capacity After Exercise Training in Elderly Heart Failure Patients With Preserved Ejection Fraction: A Randomized Exercise Trial. Arch Phys Med Rehabil. 2017 Mar;98(3):600-603. doi: 10.1016/j.apmr.2016.08.481. Epub 2016 Sep 28. PMID 27693420
- [Background] Miura Y, Fukumoto Y, Miura T, Shimada K, Asakura M, Kadokami T, Ando S, Miyata S, Sakata Y, Daida H, Matsuzaki M, Yasuda S, Kitakaze M, Shimokawa H. Impact of physical activity on cardiovascular events in patients with chronic heart failure. A multicenter prospective cohort study. Circ J. 2013;77(12):2963-72. doi: 10.1253/circj.cj-13-0746. Epub 2013 Sep 27. PMID 24077060